CLINICAL TRIAL: NCT00549861
Title: Characterization of Irreversible Myocardial Injury in Dilated Forms of Cardiomyopathies by Gadobutrol (Gadovist®)-Enhanced Cardiovascular Magnetic Resonance Imaging
Brief Title: Characterization of Irreversible Myocardial Injury in Cardiomyopathies by Contrast-enhanced CMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oliver Strohm (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Oliver Strohm, Deputy Director, University of Calgary
Organization: University of Calgary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Gadovist001
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Cardiomyopathy, Dilated; Cardiomyopathies, Secondary
Keywords: Cardiac Magnetic Resonance Imaging; Contrast agents; Gadobutrol; Fibrosis; Prognosis; Magnetic Resonance; Gadolinium
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathies; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A1 (No Intervention): CMR study for the assessment of irreversible tissue damage
  Interventions: Procedure: Cardiac Magnetic Resonance study

INTERVENTIONS:
Procedure: Cardiac Magnetic Resonance study — Cardiac MRI study

SUMMARY:
Different studies have shown that fibrosis of the heart increases the risk for a sudden death from e.g. arrhythmias. Magnetic Resonance Imaging (CMR) can easily identify even small areas of fibrosis in the heart muscle after contrast agent application (Gadolinium). With the development of faster scanners and new contrast agents, the detection of small fibrotic areas may even be improved.

In this study, we will apply dedicated T1- and T2-weighted CMR sequences before and after administration of Gadolinium-based contrast (Gadobutrol, Gadovist(r)), the study parameters will be full cardiac function, areas of edema, areas of inflammation and areas of fibrosis.

We hypothesize, that we can detect fibrotic areas in the myocardium using Gadobutrol (Gadovist (r)) better than with the commonly used Gadolinium-DTPA contrast agents. We also hypothesize, that fibrosis of the myocardium is correlated to prognosis of the patients.

DETAILED DESCRIPTION:
Dilated forms of cardiomyopathies present with left ventricular enlargement and reduced ejection fraction. Myocardial fibrosis as assessed by gradient echo sequences after contrast application ("late enhancement") has been proven to be of outstanding value for the detection of small irreversibly injured lesions and has been used to accurately characterize scarred tissue in infarcts (Kim et al, Circulation 1999), myocarditis (Mahrholdt et al., Circulation 2004), and hypertrophic cardiomyopathy (Moon et al., J Am Coll Cardiol 2004). Whereas fibrosis pattern have been described for non-ischemic cardiomyopathies (Mahrholdt et al., Eur Heart J 2005), little is known about the specific regional distribution of fibrous tissue within the group of dilated forms. McCrohon et al. have described a mid-mural and a patchy pattern in patients with global LV dysfunction and no evidence of relevant coronary artery disease (McCrohon et al., Circulation 2003). This study however, did not include right ventricular cardiomyopathy patients and patients with isolated non-compaction as two important dilated forms of cardiomyopathy.

Justification/relevance/purpose

The presence of fibrosis in dilated forms of cardiomyopathy may be predictive of progression of left ventricular dysfunction over time, as it may represent irreversible damage.

Gadobutrol will be used as the only contrast agent in this study; the significantly higher relaxivity as compared to other contrast agents will potentially allow the visualization of small, focal areas of irreversible injury in the myocardium, thus increasing sensitivity of the method to identify even localized fibrotic areas.

Objective, hypothesis

We attempt to define disease-specific patterns of extent and spatial distribution of irreversible tissue injury within the group of dilated forms of cardiomyopathies.

We hypothesize that in patients with dilated cardiomyopathies certain patterns of late enhancement can be identified, which are useful for a more specific phenotyping.

We also hypothesize that the use of Gadobutrol (Gadovist®) as the only contrast agent identifies small areas of irreversible tissue injury better than standard contrast agents and may be beneficial for diagnosing small fibrotic changes.

ELIGIBILITY:
Inclusion Criteria:

* Known cardiomyopathy (DCM, HCM, ARVC or LVNC)
* Clinical indication for contrast-enhanced Cardiac Magnetic Resonance study
* Ability to give informed consent

Exclusion Criteria:

* Any contraindication for a Magnetic Resonance Study including implanted devices, claustrophobia etc.
* Allergic reaction to Gadolinium-based contrast agents
* Known adverse reaction to Gadovist®
* Inability to give informed consent
* Known long-QT syndrome or other known conduction abnormalities
* Pregnancy or breast-feeding
* Any exclusion criteria for the administration of Gadovist® as stated in the product monograph for Warning and Precautions, e.g. Hx of allergic dispositions, or bronchial asthma; sickle cell anemia or hemoglobinopathies; renal insufficiency, with hypokalemia; convulsive states
* Conditions and concomitant medication which may prolong the QTc interval, e.g. long-QT syndrome, patients with hypokalemia, receiving Class I1 (e.g. quinidine, procainamide) or class III (amiodarone, sotalol) known antiarrhythmogenic drugs, or other medication that are known to prolong QT interval (such as cisapride, erythromycin, antipsychotic and antidepressants) - since there is a lack of clinical experience and potential risks with the concomitant use of these medication with the MRI contrast
* Patients with severe renal impairment (GFR <30mL/min)
* Patients with previous reaction to MRI and / or CT contrast media
* Patients with acute renal dysfunction due to hepato-renal syndrome or patients in the perioperative liver transplantation period
* Patients with end-stage renal disease (GFR <15mL/min/1.73m2)
* Unstable patients, e.g. from CCU / ICU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Extent and spatial distribution of irreversible tissue injury within the group of dilated forms of cardiomyopathies | within one year

SECONDARY OUTCOMES:
Use of Gadobutrol (Gadovist®) identifies small areas of irreversible tissue injury better than standard contrast agents and may be beneficial for diagnosing small fibrotic changes. | within one year

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Strohm, MD, FESC, Principal Investigator — University of Calgary
Locations (1):
- Stephenson CMR Centre at Foothills Medical Centre, University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Abdel-Aty H, Boye P, Zagrosek A, Wassmuth R, Kumar A, Messroghli D, Bock P, Dietz R, Friedrich MG, Schulz-Menger J. Diagnostic performance of cardiovascular magnetic resonance in patients with suspected acute myocarditis: comparison of different approaches. J Am Coll Cardiol. 2005 Jun 7;45(11):1815-22. doi: 10.1016/j.jacc.2004.11.069. PMID 15936612
- [Background] Jassal DS, Nomura CH, Neilan TG, Holmvang G, Fatima U, Januzzi J, Brady TJ, Cury RC. Delayed enhancement cardiac MR imaging in noncompaction of left ventricular myocardium. J Cardiovasc Magn Reson. 2006;8(3):489-91. doi: 10.1080/10976640600599502. PMID 16755837
- [Background] Maceira AM, Joshi J, Prasad SK, Moon JC, Perugini E, Harding I, Sheppard MN, Poole-Wilson PA, Hawkins PN, Pennell DJ. Cardiovascular magnetic resonance in cardiac amyloidosis. Circulation. 2005 Jan 18;111(2):186-93. doi: 10.1161/01.CIR.0000152819.97857.9D. Epub 2005 Jan 3. PMID 15630027
- [Background] Smedema JP, Snoep G, van Kroonenburgh MP, van Geuns RJ, Dassen WR, Gorgels AP, Crijns HJ. Evaluation of the accuracy of gadolinium-enhanced cardiovascular magnetic resonance in the diagnosis of cardiac sarcoidosis. J Am Coll Cardiol. 2005 May 17;45(10):1683-90. doi: 10.1016/j.jacc.2005.01.047. Epub 2005 Apr 25. PMID 15893188
- [Background] Assomull RG, Prasad SK, Lyne J, Smith G, Burman ED, Khan M, Sheppard MN, Poole-Wilson PA, Pennell DJ. Cardiovascular magnetic resonance, fibrosis, and prognosis in dilated cardiomyopathy. J Am Coll Cardiol. 2006 Nov 21;48(10):1977-85. doi: 10.1016/j.jacc.2006.07.049. Epub 2006 Oct 31. PMID 17112987
- [Background] Tandri H, Saranathan M, Rodriguez ER, Martinez C, Bomma C, Nasir K, Rosen B, Lima JA, Calkins H, Bluemke DA. Noninvasive detection of myocardial fibrosis in arrhythmogenic right ventricular cardiomyopathy using delayed-enhancement magnetic resonance imaging. J Am Coll Cardiol. 2005 Jan 4;45(1):98-103. doi: 10.1016/j.jacc.2004.09.053. PMID 15629382
- [Background] Moon JC, McKenna WJ, McCrohon JA, Elliott PM, Smith GC, Pennell DJ. Toward clinical risk assessment in hypertrophic cardiomyopathy with gadolinium cardiovascular magnetic resonance. J Am Coll Cardiol. 2003 May 7;41(9):1561-7. doi: 10.1016/s0735-1097(03)00189-x. PMID 12742298